CLINICAL TRIAL: NCT03784664
Title: Reducing Pain in Emergency Department by Using Veinous Blood Gas Instead of Arterious Blood Gas
Acronym: VEINART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Assistance Publique - Hôpitaux
Record Dates: First submitted 2018-12-12; First posted 2018-12-24 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2018-12

CONDITIONS: Acid Base Disorder
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arterial blood gas (Active Comparator)
  Interventions: Diagnostic Test: Arterial blood gas
- Veinous blood gas (Experimental)
  Interventions: Diagnostic Test: Veinous blood gas

INTERVENTIONS:
Diagnostic Test: Arterial blood gas — arterial blood sample with puncture of the radial artery
  Arms: Arterial blood gas
Diagnostic Test: Veinous blood gas — veinous blood sample using peripheral venepuncture
  Arms: Veinous blood gas

SUMMARY:
Blood gases are widely used in emergency and resuscitation services and are the key examination for exploring acid-base balance disorders (using pH, PaCO2 and HCO3 ) and gas exchange disorders (using PaO2 and PaCO2). This examination can be taken from both venous and arterial sample and its analysis depends on the type of blood sample. Currently, several studies have already shown the existence of a good correlation of pH and bicarbonates level between a venous and arterial sample. Thus, when this examination is prescribed for the purpose of highlighting and analyzing an acid-base disorder, venous blood gas is theoretically as efficient as arterial blood gas.

Due to the lack of evidence of benefit for the patient or the health care team of a venous blood gas rather than an arterial blood gas in the absence of suspicion of hypoxemia, arterial blood gas is currently the standard of care for the analysis of acid-base disorders. Indeed, among the university hospitals affiliated to the Paris Diderot University, the emergency departments carry out in their vast majority (4 of 5 E.D.) arterial blood gases. Demonstration of the superiority of veinous sample over arterial sample regarding pain could substantially modify current practices.

The investigator's main hypothesis is that, in the absence of suspicion of hypoxemia (normal oxygen saturation measured by plethysmography), the realization of a venous blood gas for the evaluation of the acid-base balance in the context of emergencies is less painful for patients, simpler for the health care team and provides sufficient biochemical information for the doctor in comparison with an arterial blood gas.

ELIGIBILITY:
Inclusion Criteria:

* necessity of blood gas analysis
* age > 18 yo
* SpO2>95% without supplemental oxygen
* no altered level of consciousness: Glasgow Coma Scale=15

Exclusion Criteria:

* Patient under guardianship or curatorship
* confusional state or patient unable to understand the protocol
* no social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Pain score: Visual Analog Scale | Immediately after blood gas sample
  Pain is self-completed by the patient using a Visual Analog Scale. Visual Analog Scale for Pain is a continuous scale comprised of a line of 100 mm grading pain intensity anchored by "no pain" (score 0) and "worst imaginable pain" (score 100)

SECONDARY OUTCOMES:
Number of attempts needed to obtain a blood gas sample | Immediately after blood gas sample
Number of different operators needed to obtain a blood gas sample | Immediately after blood gas sample
Ease of blood gas sampling procedure | Immediately after blood gas sample
  Ease of blood gas sampling procedure assessed by the operator using a four-levels likert scale ("easy","moderate","difficult" "very difficult")
Failure of the blood gas sampling procedure | Immediately after blood gas sample
  Impossibility to obtain a blood gas sample
Quality of information provided by the blood gas analysis: four levels likert scale | Immediately after having received blood gas analysis results
  Four-levels likert scale assessing doctor's satisfaction regarding the quality of gas information provided by the blood gas analysis ("very satisfied","satisfied","slightly satisfied","not satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Damien Roux, MD,PhD, Study Chair — Intensive care department, Louis Mourier hospital
Locations (4):
- France (4):
  - Hôpital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - Hôpital Lariboisière, Paris
  - Hôpital Bichat, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chauvin A, Javaud N, Ghazali A, Curac S, Altar A, Ali T, Beguin N, Bellier J, Coupier A, Delsarte L, Dreyfuss D, Kheirbek N, Oudar C, Stordeur Y, Weiss M, Gaudry S, Lambert J, Roux D. Reducing pain by using venous blood gas instead of arterial blood gas (VEINART): a multicentre randomised controlled trial. Emerg Med J. 2020 Dec;37(12):756-761. doi: 10.1136/emermed-2019-209287. Epub 2020 Aug 5. PMID 32759347